CLINICAL TRIAL: NCT02926118
Title: Continuous Glucose Monitoring During Diets That Differ in Glycemic Load
Acronym: GLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: REF-CSC-2682
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Glucose Metabolism Disorders
Keywords: Glucose; Continuous glucose monitor; Glycemic load; Dietary intervention
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low glycemic load (Experimental): Low glycemic load
  Interventions: Dietary Supplement: Low glycemic load
- High glycemic load (Experimental): High glycemic load
  Interventions: Dietary Supplement: High glycemic load

INTERVENTIONS:
Dietary Supplement: Low glycemic load — Low glycemic load diets will be consumed at breakfast, lunch and dinner for three consecutive days
  Arms: Low glycemic load
Dietary Supplement: High glycemic load — High glycemic load diets will be consumed at breakfast, lunch and dinner for three consecutive days
  Arms: High glycemic load

SUMMARY:
This study test whether a Continuous Glucose Monitor can pickup differences in glucose (in the interstitial fluid) during a dietary intervention using meals with either a high with a low glycemic load.

DETAILED DESCRIPTION:
The aim of this study is to determine the suitability of a continuous glucose monitor to detect the impact of a dietary intervention on postprandial blood glucose levels in normal, healthy, free living subjects. We will compare a dietary intervention of meals with a high glycemic load (high post-meal blood glucose) versus meals with a low glycemic load (low post-meal blood glucose) in a cross-over study. In addition, the glucose profiles obtained both via venous blood sampling and via continuous glucose monitor following a standard carbohydrate load will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy males and post-menopausal females
* Age at start of the study ≥ 50 and ≤ 70 years
* Body mass index (BMI) ≥ 25.0 and ≤ 35.0 kg/m2
* Fasting blood glucose value of subjects is ≥ 3.4 and < 6.1 mmol/L at screening
* Being used to eat three meals a day
* Having a general practitioner
* Agreeing to be informed about medically relevant personal test-results by a physician
* Accessible veins on arms as determined by examination at screening.

Exclusion Criteria:

* Having a medical conditions which might affect the study measurements (including but not limited to: diabetes type 1 and type 2, gastrointestinal disorders, gastrointestinal surgery and inflammatory diseases, as judged by the study physician
* Reported use of over-the-counter or prescribed medication or food supplements, which may interfere with study measurements as judged by the principal investigator
* Use of oral antibiotics in 40 days or less prior to the start of the study
* Reported participation in another nutritional or biomedical study 3 months before the screening or during the study
* Reported participation in night shift work 2 weeks prior to screening or during the study. Night work is defined as working between mid-night and 6.00 am
* Reported intense sporting activities > 2h/w. Intense sporting activities are defined as those activities that cause a lack of breath which limits the ability to have a normal conversation
* Reported alcohol consumption > 10 units/week (female) or > 14 units/week (male)
* Reported use of any nicotine containing products in the 6 months preceding the study and willing to abstain from use of nicotine containing products during the study itself
* Reported dietary habits: medically prescribed diet, slimming diet, vegetarian
* Reported weight loss/gain (> 3 kg) in the last 2 months before the study
* Being an employee of Unilever or research departments in NUTRIM or the Maastricht University Medical Centre (MUMC+) collaborating in this study
* Known allergy or intolerance to food products.
* Blood donation in the past 3 months

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Post prandial glucose concentration | 0 - 120 minutes after the start of each of the 3 main meals (breakfast, lunch dinner)
  Difference in glucose concentrations between the low glycemic load and the high glycemic load diet. Incremental area under the curve after the three main meals (breakfast, lunch, dinner) during both dietary interventions will be calculated. The nine post prandial periods for both low and high glycemic load diet per subject will be combined in the mixed model.

SECONDARY OUTCOMES:
Three-day glucose concentration | From start of dietary intervention until the end 3 days later
  Difference in glucose concentrations between the low and the high glycemic load diet. Total area under the curve will be compared
Day time glucose concentration | Between 07:00-22:00 h
  Difference in glucose concentrations between the low and the high glycemic load diet. Total area under the curve will be compared
Night time glucose concentration | Between 22:01-26:59 h
  Difference in glucose concentrations between the low and the high glycemic load diet. Total area under the curve will be compared
Glucose variability | From start of dietary intervention until the end 3 days later
  The Continuous Overall Net Glycemic Action (CONGA) will be calculated.
Comparison of continuous interstitial glucose with venous blood glucose | -30, -15, 15, 30, 45, 60, 90 and 120 minutes after consumption of a standard meal
  Bland-Altman plots of venous blood glucose plotted against the continuous interstitial glucose at the closest available time point. Standard meal will be 200 grams of rice consumed on the day after both the low and high glycemic load diets

OTHER OUTCOMES:
Carry over of the dietary intervention into the next day | 0 - 120 minutes after the standard meal
  Difference in glucose (in venous blood) and insulin responses to a standard meal consumed on the day after both the low and high glycemic load diets. 2-hour post prandial Incremental are under the curve for glucose and insulin in venous blood will be calculated.
Carry over as measured in venous blood versus as measured during continuous glucose monitoring | 0 - 120 minutes after the standard meal
  Compare the difference in glucose responses to the standard meal on morning after the low and the high glycemic load diet measured in venous blood with the difference as measured in using continuous blood glucose monitor. 2-hour post prandial incremental area under the curve for glucose will be calculated for both methods.
Post prandial glucose concentration during breakfast, lunch or dinner. | 0 - 120 minutes after each of the start of the meal
  Difference in post prandial glucose concentrations between the low glycemic load and the high glycemic load diet. Incremental area under the curve after each of the three main meals (breakfast, lunch, dinner) during the three-day dietary interventions will be calculated separately. The three post prandial periods for both low and high glycemic load diet per subject will be combined in separate mixed models for breakfast, a model for lunch and a model for dinner.

CONTACTS AND LOCATIONS:
Overall Officials: Mensink Ronald P, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No